CLINICAL TRIAL: NCT06110663
Title: A Phase 3, Randomized, Open-label, Multicenter Study to Assess the Efficacy and Safety of HS-10241 Combined With Almonertinib Versus Pemetrexed Combined With Platinum in Metastatic or Locally Advanced NSCLC With MET Amplification After Failure of the Prior EGFR -TKI Therapy
Brief Title: A Study of HS-10241 Combined With Almonertinib Versus Platinum-based Chemotherapy in Treatment of Advanced NSCLC With MET Amplification After Failure of EGFR-TKI Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-10241-301
Record Dates: First submitted 2023-10-24; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-10241+Almonertinib (Experimental): Experimental group (Experimental): HS-10241 combined with Almonertinib NSCLC with MET amplification after failure of EGFR-TKI treatment randomized to HS-10241 combined with Almonertinib
  Interventions: Drug: HS-10241+ Almonertinib
- Pemetrexed + Cisplatin /Carboplatin (Active Comparator): Control group (Active Comparator): Pemetrexed combined with Platinum NSCLC with MET amplification after failure of EGFR-TKI treatment randomized to standard chemotherapy treatment of platinum-based chemotherapy
  Interventions: Drug: Pemetrexed + Cisplatin /Carboplatin

INTERVENTIONS:
Drug: HS-10241+ Almonertinib — HS-10241 300mg twice daily (BID) combined with Almonertinib 110mg once daily (QD) orally, for every cycle of 21 days until disease progression or other criteria for treatment discontinuation will be met.
  Arms: HS-10241+Almonertinib
Drug: Pemetrexed + Cisplatin /Carboplatin — The standard chemotherapy treatment of cisplatin/carboplatin combined with pemetrexed for 4~6 cycles (every 3 weeks).
  Participants will continue receive pemetrexed monotherapy until disease progression or other criteria for treatment discontinuation will be met.
  Arms: Pemetrexed + Cisplatin /Carboplatin

SUMMARY:
HS-10241, an oral and highly selective MET-TKI, may contribute to overcoming common acquired MET-based resistance mechanisms following prior EGFR-TKI monotherapy. This study is conducted to evaluate the efficacy and safety of HS-10241 combined with Almonertinib versus platinum-based chemotherapy in NSCLC with MET amplification after failure of EGFR-TKI treatment.

DETAILED DESCRIPTION:
This is a phase 3, randomized, open-label, multicenter study to evaluate the efficacy and safety of HS-10241 in combination with Almonertinib versus platinum-based chemotherapy in patients with MET-amplified locally advanced or metastatic NSCLC who have progressed after prior EGFR-TKI therapy.

All eligible patients were randomly assigned to experimental group (HS-10241 combined with Almonertinib) or control group (pemetrexed combined with platinum) at a ratio of 1:1. Patients in experimental group will receive HS-10241 300mg twice daily (BID) combined with Almonertinib 110mg once daily (QD) orally and will continue treatment until disease progression or other criteria for treatment discontinuation will be met. Patients in control group will receive the standard chemotherapy treatment of cisplatin/carboplatin combined with pemetrexed for 4~6 cycles. Participants will continue receive pemetrexed monotherapy until disease progression or other criteria for treatment discontinuation will be met. The efficacy and safety of the two groups will be evaluated after follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged more than or equal to (≥) 18 years.
2. Patients histologically or cytologically confirmed with locally advanced or metastatic NSCLC.
3. Patients have previously received EGFR TKI treatment and had intolerance or disease progression by imaging recorded. Chemotherapy as systematic therapy is limited to no more than one prior line. Before randomization, all patients must provide imaging evidence of disease progression during or after the last treatment period. The patients are required to provide tumor biopsy tissue (required) and blood samples (optional) of disease progression after the last treatment of EGFR TKI, confirmed by central laboratory that there are EGFR sensitive mutations (deletion of exon 19 or L858R mutation) and T790M status (negative or positive) in tumor tissues and/or blood samples. Meanwhile, the tumor tissue should be c-MET positive confirmed by the central laboratory.
4. According to Recist1.1, at least 1 target lesion that should be measurable lesions without local treatment like irradiation or with definite progression after local treatment and can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes, which must have short axis ≥ 15mm)
5. ECOG performance status of 0-1with no deterioration within 2 weeks before enrollment.
6. Estimated life expectancy ≥three months.
7. Females of child bearing age should adapt adequate contraceptive measures and should not be breastfeeding from the signing of informed consent to 6 months after the last treatment of the study. Male patients should be willing to use barrier contraception (i.e., condoms) from the signing of informed consent to 6 months after the last treatment of the study.
8. Females must have a negative pregnancy test in 7 days prior to the date of randomization if of childbearing potential or must have evidence of non-childbearing potential by fulfilling any one of the criteria.
9. Signed and dated Informed Consent Form.

Exclusion Criteria:

1. Treatment with any of the following:

   1. Previous or current treatment with drugs targeting the c-MET/HGF pathway.
   2. Previous or under treatment with pemetrexed and platinum.
   3. Any cytotoxic chemotherapy, investigational agents, antitumor traditional Chinese Medicine and any other anticancer drugs for the treatment of advanced NSCLC within 14 days before the date of randomization; or requiring treatment with these drugs during the study.
   4. Any antitumor monoclonal antibody therapy within 28 days before the date of randomization.
   5. Local radiotherapy within 2 weeks of the date of randomization; receiving radiation to > 30% of the bone marrow or with a wide field of radiation within 4 weeks before the date of randomization.
   6. Spinal cord compression or brain metastases (except for that being asymptomatic and stable for at least 4 weeks, not requiring steroids for at least 2 weeks prior to start of study treatment and with no obvious edema around the tumor focus by imaging examination).
   7. Currently receiving drugs known to prolong QT interval or may cause torsade de pointe; or requiring treatment with these drugs during the study.
2. Any unresolved toxicities from prior therapy greater than Grade 2 according to Common Terminology Criteria for Adverse Events (CTCAE) 5.0 with the exception of alopecia or neurotoxicity.
3. History of other primary malignancies.
4. Inadequate bone marrow reserve or organ function, as demonstrated by any of the following laboratory values:

   1. Absolute neutrophil count (ANC) <1.5×109 / L
   2. Platelet count <90×109 / L
   3. Hemoglobin <90 g/L
   4. Total bilirubin (TBL) > 1.5 × ULN or > 3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases.
   5. One or both of Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) > 2.5 × upper limit of normal (ULN) or > 5 × ULN in the presence of liver metastases.
   6. Creatinine > 1.5 × ULN concurrent with creatinine clearance < 50 mL/min; confirmation of creatinine clearance is only required when creatinine is > 1.5 × ULN.
   7. International normalized ratio (INR) > 1.5, and partially activated prothrombin time (APTT) > 1.5 × ULN.
   8. Serum albumin (ALB) < 28 g/L
5. Any of the following cardiac criteria:

   1. Resting corrected QT interval (QTc) > 470 ms obtained from electrocardiogram (ECG), using the screening clinic's ECG machine and Fridericia's formula for QT interval correction (QTcF).
   2. Left ventricular ejection fraction (LVEF) ≤ 50%.
6. Severe, uncontrolled or active cardiovascular diseases.
7. Diabetes ketoacidosis or hyperglycemia hypertonic occurring within 6 months before the date of randomization, or the glycosylated hemoglobin value ≥ 7.5% in the screening period.
8. Severe or poorly controlled hypertension.
9. Hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh Grade B or more severe cirrhosis.
10. Other moderate or severe lung diseases that may interfere with the detection or treatment of drug-related pulmonary toxicity or may seriously affect respiratory function.
11. Women who are breastfeeding or pregnant or planned to be pregnant during the study period.
12. History of hypersensitivity to any active or inactive ingredient of HS-10241/Almonertinib/ cisplatin/carboplatin/pemetrexed or to drugs with a similar chemical structure or class to HS-10241/Almonertinib/cisplatin/carboplatin/pemetrexed.
13. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
14. Any disease or condition that, in the opinion of the investigator, would compromise the safety of the patient or interfere with study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) evaluated by Independent Review Committee (IRC) | From the date of randomization to the earliest date of the first objective documentation of radiographic disease progression or death due to any cause, assessed up to 24 months
  Progression of tumor was assessed by RECIST 1.1 thereby to evaluate progression free survival. Progression-free survival was deﬁned as the time from date of randomization until the documentation of objective disease progression (PD) or death from any cause in the absence of progression (whichever occurred first), regardless of whether they subsequently received non-study anti-cancer therapy.

SECONDARY OUTCOMES:
Objective response rate (ORR) evaluated by Independent Review Committee (IRC) | From the date of randomization to disease progression or date of death from any cause, whichever comes first, assessed up to 24 months.
  ORR was defined as the percentage of patients with a complete response (CR) or partial response (PR) that was confirmed at a subsequent scan at least 4 weeks later, as assessed according to RECIST version 1.1
Disease control rate (DCR) evaluated by Independent Review Committee (IRC) | From the date of randomization to disease progression or date of death from any cause, whichever comes first, assessed up to 24 months.
  Objective response was assessed by RECIST 1.1 thereby to evaluate disease control rate. Disease control was deﬁned as the percentage of patients who have a best overall response (confirmed CR, PR, or stable disease for at least 5 weeks)
Duration of response (DoR) evaluated by Independent Review Committee (IRC) | From the date of randomization to disease progression or date of death from any cause, whichever comes first, assessed up to 24 months.
  Duration of response assessed by RECIST 1.1. Duration of response was defined as the time from when the criteria for CR or PR were first met to the occurrence of an objective disease progression (PD) or death.
Overall survival (OS) | From the date of randomization up to the date of date of death from any cause，assessed up to 24 months.
  OS was defined as time from randomization until the date of death due to any cause.
Incidence and severity of treatment-emergent adverse events | From the date of randomization until 28 days after the last dose
  Assessed by number and severity of adverse events as recorded on the case report form NCI CTCAE v5.0.